CLINICAL TRIAL: NCT05003349
Title: Additional Effect of Pain Neuroscience Education, Motor Imagery and Action Observation in Patients With Chronic Temporomandibular Disorders. A Randomized Controlled Trial
Brief Title: Pain Neuroscience Education, Motor Imagery and Action Observation in Patients With Chronic Temporomandibular Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Mauro Barone, PT, University of Gran Rosario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNE, MI and AO in TMD
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: TMD
Keywords: Pain Neuroscience Education; Motor Imagery; Action Observation; Exercises; Occlusal Splint
MeSH Terms: conditions — Motor Activity | interventions — Occlusal Splints; Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Occlusal Splint (OS) + Pain Neuroscience Education (PNE) + Motor Imagery (MI) + Action Observation (AO) + Jaw and Neck Exercises (JNE) All participants in this arm will receive OS (they must use every night during the study) and will receive physiotherapy treatment including PNE, MI, AO and JNE, in 2 sessions per week, each lasting 60 minutes, during 5 weeks. For PNE a power-point presentation with metaphors, images and videos will be employed. For the MI, the participants will be asked to judge the laterality of different cervical images presented on the screen of a cell phone. The laterality task will be executed using an application called Recognize Neck, developed by the NOI group. The AO will be carried out using videos of mandibular and cervical exercises. The JNE program will be performed 3 sets of 10 repetitions. The exercises will be executed with a total time per session of 20 minutes, initially at the clinic and later at home.
  Interventions: Other: Occlusal Splint (OS).; Other: Pain Neuroscience Education (PNE).; Other: Motor Imagery (MI).; Other: Action Observation (AO).; Other: Jaw and Neck Exercises (JNE)
- Active comparator (Active Comparator): Occlusal Splint (OS) + Counselling + Jaw and Neck Exercises (JNE). All participants in this arm will receive OS and will receive physiotherapy treatment including Counselling and JNE, in 2 sessions per week, each lasting 40 minutes, during 5 weeks. The JNE will be administered in the same way as in the other arm of the study.
  Counselling include education about the anatomical, biomechanical and psychosocial factors relationed with temporomandibular disorders, guidance regarding the parafunction jaw activities for eg will be taught the resting postural position of the mandible (teeth apart, lips slightly touching and tongue not pushing against the teeth).
  Interventions: Other: Occlusal Splint (OS).; Other: Jaw and Neck Exercises (JNE); Other: Counselling.

INTERVENTIONS:
Other: Occlusal Splint (OS). — OS will be made of heat-cured acrylic by the same specialized dentist. These intraoral devices will be flate, rigid, will cover the entire dental arch, and will have the lowest possible height. The perimeter of the splint will have at least 11 dental contacts, light, symmetrical and pinpoint as possible. The patients will be instructed to use the splint every night during the study Two supervisions will be carried out 30 and 60 days after the use of the OS, in order to stabilize the contact points.
Other: Pain Neuroscience Education (PNE). — A power point presentation with metaphors and animated videos will be used. The PNE will be held in 10 sessions of 20 minutes each. The intervention will be developed using content according to the book "Explain Pain" and the web page www.retrainpain.org.
  Arms: Experimental group
Other: Motor Imagery (MI). — The participants will have to judge the laterality of different cervical images presented on the screen of a cell phone. The laterality task will be executed using an application called Recognize Neck, developed by the NOI group. The procedure will begin with a familiarization test with the "Basic" level followed by a laterality discrimination task. It will be performed using 20 images, with 5 seconds for each image, beginning with the "Vanilla" program and progressively increasing the difficulty using the "Context" and "Abstract" programs. The estimated time to complete the task will be about 10 minutes per session.
  Arms: Experimental group
Other: Action Observation (AO). — The patients will see videos showing the jaw and cervical exercises with the same series and repetitions that they will actively perform in the session. Therefore, the training of the action observation will be carried out dynamically. The patient will be asked to think and visualize the movement that he/she will have to perform later. It is estimated 10 minutes per session for the AO.
  Arms: Experimental group
Other: Jaw and Neck Exercises (JNE) — A jaw and neck exercise program will be carried out in 3 series of 10 repetitions per session will be planned with 1minute rest between exercise. The exercises will be executed with a total time per session of 20 minutes, initially in the clinic and later at home. In the clinic, verbal and tactile instructions will be provided for the correct execution of the exercises and later they will be sent through WhatsApp and / or mail to perform them at home.
Other: Counselling. — Counselling include education about the anatomical, biomechanical and psychosocial factors relationed with temporomandibular disorders, guidance regarding the parafunction jaw activities for eg will be taught the resting postural position of the mandible (teeth apart, lips slightly touching and tongue not pushing against the teeth).
  Arms: Active comparator

SUMMARY:
The objective of this study will be to verify the additional effect of Pain Neuroscience Education, Motor Imagery and Action Observation on primary outcomes pain intensity and craniofacial pain and disability in patients with chronic temporomandibular disorders (TMD). The secondary outcomes will be pressure pain threshold, temporal summation, conditioned pain modulation, central sensibilization, pain catastrophizing, kinesiophobia. This study will be a doble-blinded randomized clinical trial comprising a sample of 50 participants with orofacial pain of both genders and aged between 18 and 60 years. Subjects will undergo a screening process to identify those presenting a diagnosis of painful TMD confirmed by the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD), and then they will be randomized into two groups (G1: Occlusal Splint, Counselling and Jaw and Neck Exercises vs. (G2: Occlusal Splint, Jaw and Neck Exercises plus Pain Neuroscience Education, Motor Imagery and Action Observation). These volunteers will be recruited from the Alisos Group Dentistry Clinic and University of Gran Rosario, (Rosario, Argentina). All patients will wear an occlusal splint designed by dentists. The interventions will be administered twice a week for 5 weeks by a single therapist. Subsequently, patients will be given instructions to perform the exercises at home for 5 weeks. Primary and secondary outcomes will be measured at baseline, 6 weeks and 12 weeks, and at 3 months after the end of treatment (follow-up). All the evaluations will be performed by a blinded physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of painful TMD using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
* A history of orofacial pain during at least three months prior to the study
* Age ranging between 18 to 65 years, both genders.

Exclusion Criteria:

• Patients with neurological disorders (neuropathic pain or neurodegenerative disease), whiplash associated disorders, specific neck pain (radicular pain), recent dental or physical therapy. If patients are taking medication to relieve pain during the study, they will be encouraged to report it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity. | At baseline, then at six, twelve weeks, and 3 months follow-up.
  The Numerical Pain Rating Scale (NPRS) will be used to assess pain intensity. This scale consists in a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change in Craneofacial pain and disability inventory. | At baseline, then at six, twelve weeks, and 3 months follow-up.
  The Craneofacial pain and disability inventory (CF-PDI) is a self-administered questionnaire that has been designed to obtain information on how pain in the orofacial region affects the patient's daily life. It consists of 21 items, with the final score ranging from 0 to 63 points. Each question is scored on a 4-point ordinal scale, ranging from 0 to 3. A higher score reflects higher pain and disability levels.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold. | At baseline, then at six, twelve weeks, and 3 months follow-up
  The Pressure Pain Threshold (PPT) will be measured through a pressure algometer in 3 different sites; 1) Anterior temporalis muscle, 2) upper trapezius muscle and 3) thenar eminence (non-dominant hand). At each site, 3 measurements will be made with an interval of 30 seconds, and the mean will be registered. To determine the PPT, the pressure will be increased at a rate of approximately 1 kg/second and patients will be asked to raise their arm the moment the pressure begins to change to a sensation of pain, at which point, the evaluator will stop pressing. PPT values will be expressed in kg/cm2.
Change in Temporal Summation. | At baseline, then at six, twelve weeks, and 3 months follow-up
  Temporal Summation (TS) will be induced using a pressure algometer. For TS, 10 consecutive pressure pulses will be elicited using the PPT (obtained before). For each pulse of the TS procedure, the pressure will increase at a rate of 1 kg/second until the PPT is reached, where it will remain for one second before being released. The pressure pulses will be repeatedly performed with an interval between stimuli of one second. Participants will be instructed to assess the pain intensity of the first and tenth pressure pulses according to the NPRS. The TS score will be obtained by subtracting the first NPRS score from the last score. The higher the TS score, the more efficient nociceptive signaling for the brain.
Change in Conditioned Pain Modulation. | At baseline, then at six, twelve weeks, and 3 months follow-up
  For the Conditioned Pain Modulation (CPM) a occlusion cuff will be used as a conditioning stimulus. The cuff will be inflated in the non-dominant arm at approximately 20 mm Hg/second until the subjects report experiencing pain at a value of 5/10 using the NPRS, when inflation will stop. Subjects will adapt to the stimulus for 30 seconds, and the first PPT measurement will be performed. Then, the cuff will then be deflated and 1 minute later the second PPT measurement will be taken.
Change in Central Sensibilization Inventory. | At baseline, then at six, twelve weeks, and 3 months follow-up
  The Central Sensibilization Inventory (CSI) is a self-report outcome measure that consists of two parts. Part A consists of 25 statements where the participant must answer how often he/she experience each symptom. Individual items are scored from "0" (never) to "4" (always), resulting in a total score range for all 25 items from "0" to "100". Part B asks if the participant have been previously diagnosed by a doctor for some diseases (YES/NO). Part B of the CSI is for information only and is not qualified. A score of more than 40 indicates the presence of central sensitization.
Change in Pain Catastrophizing Scale | At baseline, then at six, twelve weeks, and 3 months follow-up
  The Pain Catastrophizing scale (PCS) is a 13-items instrument that ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points being (0) not at all and, (4) all the time. A total score (ranging from 0 to 52) is obtained, along with three subscale scores that assess rumination, magnification, and helplessness. A higher total PCS score of 30 represents a clinically relevant level of catastrophizing.
Change in Spanish version of the Tampa Scale of Kinesiophobia for Temporomandibular. Disorders | At baseline, then at six, twelve weeks, and 3 months follow-up
  The Spanish version of the Tampa Scale of Kinesiophobia for Temporomandibular Disorders (TSK-TMD-S) consists of 10 items formulated positively and distributed in 2 subscales as follows: (1) somatic approach (items 1, 2, 3, 4 and 10) and (2) avoidance of activities (items 5 to 9). The total score can range from 10 to 40 (somatic focus, 5-20; avoidance of activity, 5-20), with higher scores indicating an increased fear of jaw movement and re-injury. The cut-off point to consider kinesiophobia is 23 points.
Change in Home exercise adherence | Between the sixth and twelfth week (once per week)
  To assess adherence to home exercise, a google form will be sent weekly to the volunteers. It will consist of questions related to the number of times patients performed the exercises during the week and to the difficulties they encountered. Adherence to exercises will be expressed as a percentage [(number of exercise sessions performed / number of exercise sessions prescribed) X100].

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: No